CLINICAL TRIAL: NCT00118274
Title: A Multicenter Trial to Evaluate the Effects of Administration of Cyclophosphamide and Melanoma-Derived Helper Peptides on the Immunogenicity of a Class I MHC-Restricted Peptide-Based Vaccine in Participants With Resected Melanoma
Brief Title: Vaccine Therapy With or Without Cyclophosphamide in Treating Patients Who Have Undergone Surgery for Stage II, Stage III, or Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Professor of Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11491; UVACC-34104; UVACC-MEL-44; UVACC-GCRC-CLS013; UVACC-HITC-02620; MDA-2005-0070
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — incomplete Freund's adjuvant; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I (Experimental): Patients receive vaccine comprising multi-epitope melanoma peptides, tetanus toxoid helper peptide emulsified in Montanide ISA-51 intradermally and subcutaneously on days 1, 8, 15, 29, 36, 43, 85, 183, 274, and 365.
  Interventions: Biological: incomplete Freund's adjuvant; Biological: multi-epitope melanoma peptide vaccine; Biological: tetanus toxoid helper peptide
- Arm II (Experimental): Patients receive cyclophosphamide IV over 30-60 minutes on day -4. Patients then receive vaccine comprising multi-epitope melanoma peptides, tetanus toxoid helper peptide emulsified in Montanide ISA-51 intradermally and subcutaneously on days 1, 8, 15, 29, 36, 43, 85, 183, 274, and 365.
  Interventions: Biological: incomplete Freund's adjuvant; Biological: multi-epitope melanoma peptide vaccine; Biological: tetanus toxoid helper peptide; Drug: cyclophosphamide
- Arm III (Experimental): Patients receive vaccine comprising melanoma peptides and multi-epitope melanoma helper peptides emulsified in Montanide ISA-51 intradermally and subcutaneously on days 1, 8, 15, 29, 36, 43, 85, 183, 274, and 365.
  Interventions: Biological: incomplete Freund's adjuvant; Biological: melanoma helper peptide vaccine; Biological: multi-epitope melanoma peptide vaccine
- Arm IV (Experimental): Patients receive cyclophosphamide IV over 30-60 minutes on day -4. Patients then receive vaccine comprising melanoma peptides and multi-epitope melanoma helper peptides emulsified in Montanide ISA-51 intradermally and subcutaneously on days 1, 8, 15, 29, 36, 43, 85, 183, 274, and 365.
  Interventions: Biological: incomplete Freund's adjuvant; Biological: melanoma helper peptide vaccine; Biological: multi-epitope melanoma peptide vaccine; Drug: cyclophosphamide

INTERVENTIONS:
Biological: incomplete Freund's adjuvant — Given intradermally and subcutaneously
Biological: melanoma helper peptide vaccine — Given intradermally and subcutaneously
  Arms: Arm III; Arm IV
Biological: multi-epitope melanoma peptide vaccine — Given intradermally and subcutaneously
Biological: tetanus toxoid helper peptide — Given intradermally and subcutaneously
  Arms: Arm I; Arm II
Drug: cyclophosphamide — Given IV
  Arms: Arm II; Arm IV

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Cyclophosphamide may also stimulate the immune system in different ways and stop tumor cells from growing. Giving vaccine therapy together with cyclophosphamide after surgery may cause a stronger immune response to kill any remaining tumor cells. It may also prevent or delay the recurrence of melanoma.

PURPOSE: This randomized phase I/II trial is studying the side effects of vaccine therapy when given with or without cyclophosphamide and to see how well they work in treating patients who have undergone surgery for stage II, stage III, or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of adjuvant vaccine therapy comprising multi-epitope melanoma peptides (MP) and multi-epitope melanoma helper peptides (MHP) emulsified in Montanide ISA-51 in patients with resected stage IIB-IV melanoma.
* Determine the safety of administering cyclophosphamide before vaccination in these patients.
* Compare the magnitude of immune response against vaccination comprising MP in combination with either MHP or tetanus toxoid helper peptide (TET) emulsified in Montanide ISA-51 with vs without cyclophosphamide in these patients.

Secondary

* Compare the response rate and persistence of immune responses in patients treated with these regimens.
* Compare the magnitude of immune response against vaccination comprising TET or MHP with vs without cyclophosphamide in these patients.
* Compare the response rate and persistence of immune response against vaccination comprising TET or MHP with vs without cyclophosphamide in these patients.
* Determine the delayed-type hypersensitivity response to the peptide components of these vaccines in these patients.
* Compare, preliminarily, disease-free survival of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to HLA-type (HLA-A1 positive vs HLA-A2 positive, HLA-A1 negative, or -A3 negative vs HLA-A3 positive, or -A1 negative) and participating center (University of Virginia [UVA] vs non-UVA). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive vaccine comprising multi-epitope melanoma peptides (MP) and tetanus toxoid helper peptide emulsified in Montanide ISA-51 intradermally (ID) and subcutaneously (SC) on days 1, 8, 15, 29, 36, 43, 85, 183, 274, and 365.
* Arm II: Patients receive cyclophosphamide IV over 30-60 minutes on day -4. Patients then receive vaccine as in arm I.
* Arm III: Patients receive vaccine comprising MP and multi-epitope melanoma helper peptides emulsified in Montanide ISA-51 ID and SC on days 1, 8, 15, 29, 36, 43, 85, 183, 274, and 365.
* Arm IV: Patients receive cyclophosphamide as in arm II. Patients then receive vaccine as in arm III.

Treatment in all arms continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 173 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed melanoma

  * Cutaneous, mucosal, or primary melanoma
  * Stage IIB-IV disease
* Has undergone surgical resection or stereotactic radiosurgery for malignant melanoma ≥ 1 week but ≤ 6 months ago

  * No clinical or radiological evidence of disease after surgical resection or stereotactic radiosurgery by chest x-ray or CT scan*, abdominal and pelvic CT scan*, and head CT scan or MRI NOTE: *Positron emission tomography scan/CT fusion scan may replace scans of the chest, abdomen, and pelvis
* Must have ≥ 2 intact (undissected) axillary and/or inguinal lymph node basins
* HLA-A1, -A2, or -A3 positive AND HLA-DR1, -DR4, -DR11, -DR13, or -DR15 positive
* Ineligible for OR refused interferon
* No ocular melanoma
* Brain metastases allowed provided all of the following criteria are met:

  * No more than 3 total brain metastases
  * Each metastasis ≤ 2 cm in diameter at the time of study entry
  * Each metastasis was completely removed by surgery or treated with stereotactic radiosurgery
  * No evidence of brain metastasis progression since the most recent treatment

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9 g/dL

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.5 times ULN
* Lactic dehydrogenase ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Hepatitis C negative

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No New York Heart Association class III or IV heart disease

Immunologic

* HIV negative
* No known or suspected allergy to any component of the study vaccines
* No autoimmune disorder with visceral involvement
* No prior or active autoimmune disorder requiring cytotoxic or immunosuppressive therapy
* The following immunologic conditions are allowed:

  * Laboratory evidence of autoimmune disease (e.g., positive anti-nuclear antibody titer) without symptoms
  * Clinical evidence of vitiligo
  * Other forms of depigmenting illness
  * Mild arthritis requiring non-steroidal anti-inflammatory drugs

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Weight ≥ 110 lbs
* No uncontrolled diabetes

  * Hemoglobin A1C < 7%
* No medical contraindication or potential problem that would preclude study compliance
* No other malignancy except squamous cell or basal cell skin cancer without known metastasis, carcinoma in situ of the breast (ductal or lobular) or cervix, or other successfully treated cancer without distant metastasis with no evidence of recurrence or metastasis for > 5 years
* No known active addiction to alcohol or drugs
* No recent (within the past year) or ongoing illicit IV drug use

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior vaccination with any of the synthetic peptides used in this study

  * Prior vaccinations (containing agents other than the synthetic peptides used in this study) that resulted in recurrent disease during or after vaccine administration allowed provided the last vaccination was administered more than 12 weeks ago
* More than 4 weeks since prior and no concurrent interferon (e.g., Intron-A®), interleukins (e.g., Proleukin®), or growth factors (e.g., Procrit®, Aranesp®, or Neulasta®)
* More than 4 weeks since prior and no concurrent allergy desensitization injections
* No influenza vaccines for at least 2 weeks before or after study vaccine administration

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No concurrent chemotherapy, including nitrosoureas

Endocrine therapy

* More than 4 weeks since prior and no concurrent oral or parenteral corticosteroids
* No prior or concurrent inhaled steroids (e.g., Advair®, Flovent®, or Azmacort®)
* Prior or concurrent topical corticosteroids allowed

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since other prior and no concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* More than 4 weeks since prior and no other concurrent investigational agents
* More than 30 days since prior and no concurrent participation in another clinical study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2005-03 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Slingluff, MD, Principal Investigator — University of Virginia
Locations (3):
- United States (3):
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia

REFERENCES:
- [Result] Slingluff CL Jr, Petroni GR, Chianese-Bullock KA, Smolkin ME, Ross MI, Haas NB, von Mehren M, Grosh WW. Randomized multicenter trial of the effects of melanoma-associated helper peptides and cyclophosphamide on the immunogenicity of a multipeptide melanoma vaccine. J Clin Oncol. 2011 Jul 20;29(21):2924-32. doi: 10.1200/JCO.2010.33.8053. Epub 2011 Jun 20. PMID 21690475

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Started | 41 | 43 | 42 | 44
Completed | 21 | 21 | 25 | 29
Not Completed | 20 | 22 | 17 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Arm III | Arm IV | Total
Number analyzed (Participants) | 41 | 43 | 42 | 44 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 33 | 32 | 125
  >=65 years | 11 | 13 | 9 | 12 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 13 | 13 | 56
  Male | 28 | 26 | 29 | 31 | 114

OUTCOME MEASURES:

1. Primary Outcome: Safety of the Peptide Vaccines
Description: Number of participants with dose-limiting toxicities
Time Frame: 30 days after receiving the last dose of study drug, up to week 52
Population: Intent to treat population including 167 eligible and 3 ineligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 41 | 43 | 42 | 44
Participants | 4 | 7 | 2 | 1

2. Secondary Outcome: Immunogenicity (CD8+ T Cell Response to 12 Melanoma Peptides, 12MP) as Measured by Elispot Assay, up to Day 50
Description: The primary end point was the maximum cumulative circulating CD8+ T cell response to 12 melanoma peptides (12MP) measured by ELISpot assay over the first six vaccines (to day 50).
Time Frame: 50 days
Population: All eligible participants, total = 167.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 41 | 41 | 42 | 43
Participants | 32 | 29 | 8 | 12

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II | Arm III | Arm IV
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/43 | 0/42 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43 | 0/42 | 0/44
Other Adverse Events (participants affected / at risk) | 41/41 | 43/43 | 41/42 | 44/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=41) | Arm II (N=43) | Arm III (N=42) | Arm IV (N=44)
Autoimmune reaction (Immune system disorders) | 0 | 5 | 3 | 2
Rhinitis (Immune system disorders) | 8 | 14 | 14 | 6
Hemoglobin (Blood and lymphatic system disorders) | 18 | 15 | 8 | 16 — decreased hemoglobin
Leukocytes (Blood and lymphatic system disorders) | 8 | 6 | 5 | 11
Lymphopenia (Blood and lymphatic system disorders) | 9 | 8 | 4 | 7
neutrophils (Blood and lymphatic system disorders) | 2 | 4 | 4 | 2
platelets (Blood and lymphatic system disorders) | 1 | 0 | 3 | 1
Fatigue (General disorders) | 22 | 38 | 28 | 30
Fever (General disorders) | 15 | 28 | 14 | 14
Rigors/chills (General disorders) | 26 | 33 | 17 | 18
Sweating (General disorders) | 16 | 25 | 16 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 2
Flushing (Skin and subcutaneous tissue disorders) | 8 | 9 | 10 | 6
hypopigmentation (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 2 — vitiligo
injection site reaction (Skin and subcutaneous tissue disorders) | 40 | 43 | 38 | 43
Pruritis (Skin and subcutaneous tissue disorders) | 5 | 8 | 6 | 8
Rash (Skin and subcutaneous tissue disorders) | 9 | 13 | 6 | 7
Ulceration (Skin and subcutaneous tissue disorders) | 12 | 19 | 3 | 10 — ulceration at vaccine site
Anorexia (Gastrointestinal disorders) | 14 | 22 | 14 | 12
Constipation (Gastrointestinal disorders) | 1 | 4 | 2 | 5
Diarrhea (Gastrointestinal disorders) | 13 | 13 | 11 | 11
Mucositis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 7 | 6 | 5 | 3
Nausea (Gastrointestinal disorders) | 17 | 24 | 15 | 25
Vomiting (Gastrointestinal disorders) | 5 | 10 | 2 | 7
Edema: limb (Blood and lymphatic system disorders) | 2 | 3 | 4 | 0
ALT (Hepatobiliary disorders) | 1 | 0 | 1 | 3
AST (Hepatobiliary disorders) | 4 | 2 | 4 | 4
Bilirubin (Hepatobiliary disorders) | 2 | 3 | 4 | 2
Hypercalcemia (Investigations) | 0 | 0 | 3 | 1
Hyperglycemia (Investigations) | 10 | 21 | 12 | 16
Hyperkalemia (Investigations) | 9 | 9 | 7 | 6
Hypocalcemia (Investigations) | 0 | 3 | 0 | 0
Hypoglycemia (Investigations) | 2 | 3 | 4 | 5
Hypokalemia (Investigations) | 1 | 3 | 0 | 3
Hyponatremia (Investigations) | 1 | 4 | 1 | 4
Dizziness (Nervous system disorders) | 12 | 11 | 8 | 9
Mood alteration - agitation (Psychiatric disorders) | 2 | 0 | 3 | 4
Mood alteration - anxiety (Psychiatric disorders) | 2 | 2 | 3 | 0
Mood alteration - depression (Psychiatric disorders) | 3 | 2 | 1 | 1
Pain - extremity - limb (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 0
Pain - headache (General disorders) | 24 | 25 | 21 | 16
Pain - joint (Musculoskeletal and connective tissue disorders) | 16 | 14 | 12 | 14
Pain - muscle (Musculoskeletal and connective tissue disorders) | 21 | 22 | 12 | 12
Pain - other (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 4
Pain - throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 9 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 14 | 15 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 5 | 4
Nasal/paranasal reaction (Respiratory, thoracic and mediastinal disorders) | 10 | 14 | 11 | 11
Flu-like syndrome (General disorders) | 10 | 13 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes